CLINICAL TRIAL: NCT05002907
Title: Epidemiology of Hepatitis B, C and D and HIV Along the Maroni River Bordering French Guiana and Suriname (MaHeVi)
Acronym: MaHeVi
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Foundation for Scientific Research Suriname (SWOS) Paramaribo, Suriname (Unknown)
Responsible Party: Sponsor
Other Study IDs: MaHeVi
Record Dates: First submitted 2021-07-27; First posted 2021-08-12 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis B; Hepatitis C; Hepatitis D; HIV Infections; Prevalence; Epidemiology
Keywords: Epidemiology; Prevalence; Hepatitis B; Hepatitis C; Hepatitis D; HIV Infections; Phylogenetic; Molecular Biology
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Hepatitis D; HIV Infections | interventions — Surveys and Questionnaires; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Capillary blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General adult population living along the Maroni River in French Guiana and Suriname: General adult population living along the Maroni River in French Guiana and Suriname, upstream from Apatou. All adults (men and women) 18 years or older of both sexes will be able to participate in the study, in French Guiana and Suriname. Participation will be based on volunteering and signing informed consent. The acceptability and diversity of recruitment will be improved by seeking community support through community leaders and local associations and through appropriate communication (radio spots, posters in health centers and public establishments) before the survey .
  Interventions: Other: Questionnaire; Other: Biocollection; Other: Delivery of results; Other: Results and advices on transmission prevention methods; Other: Confirmation of results on a blood test (In the event of a positive result); Other: Information for care; Other: Monitoring and treatment

INTERVENTIONS:
Other: Questionnaire — After signing the informed consent sheet, a standardized face-to-face questionnaire will be conducted by the doctor, nurse or coordinator to collect socio-demographic data, lifestyle data, sex life and other potential risk factors and knowledge about viral hepatitis.
Other: Biocollection — After answering the questionnaire, the nurse or the doctor will take a sample of capillary blood from the fingertip on the side of the distal phalanx of a middle or ring finger. The puncture site will be prepared by warming and massage to optimize blood flow and disinfected with a disposable 70% alcohol wipe. After drying, the puncture will be performed using a single use safety lancet. A total of 7 capillary blood spotswill be collected and deposited on the filter paper (each spot is about 50µL of capillary blood), 5 for the study and 2 for the biological collection.
Other: Delivery of results — After receiving the individual biological analysis results, in coded form (results only identified by the anonymity number), at the investigation center and lifting the anonymity by the coordinator of the study in each study center (in Cayenne or Paramaribo depending the country where the inclusion took place) with the help of the correspondance list, the participants' results will be delivered to the referral doctor of each health centre and the infectious disease specialist responsible for each area of inclusion. All positive participants will be contacted if they do not spontaneously come to retrieve their results (within approximately 1 month after result's availability), and invited to come to the health centre to retrieve their results individually and be oriented towards the heathcare circuit.
Other: Results and advices on transmission prevention methods — The results will be revealed by the health centre's doctor/infectiologist, individually and confidentially, with an explanation of the results and advices on transmission prevention methods.Non-immunized patients against HBV will be offered a status determination (Anti-HBs Ab quantification on whole blood sample) and if necessary a catch-up vaccination according to the national immunization schedule.
Other: Confirmation of results on a blood test (In the event of a positive result) — In case of a positive result, the doctor will explain the need to confirm these results on a blood test, prescribe the initial assessment and take an appointment with the infectious disease specialist. He will guide the patient towards accompaniment for the opening of medical coverage rights if necessary and support by an association if desired.
Other: Information for care — A document with all contact information for a comprehensive and specialized care (professionals and associations for access to medical coverage and support, associations proposing support, general practitioners and specialists) will be given to positive participants. Patient monitoring and treatment will be carried out according to the national guidelines in each country.
Other: Monitoring and treatment — Consequently, all positive participants will be able to be monitored and treated by a specialist of the disease. They will give post-test counselling and will conduct patient follow-up and treatment according to the usual standards of care of each country.

SUMMARY:
MaHeVi is a multicenter, cross-sectional, population-based study which will include 2500 adults in the health care centers / missions located on the 2 sides of the Maroni River. All major inhabitants of the river border between French Guiana and Suriname may participate, after an extensive communication campaign.The main objective is to estimate the prevalence and status of infection with hepatitis B (HBV), hepatitis C (HCV), D (VHD) and HIV in the general adult population of the Maroni River, border between French Guiana and Suriname. After signing the informed consent and pre-test counseling, capillary blood will be collected on blotting paper. Participants will be interviewed on infection risk factors. Positivity for HBsAg, total anti-HBcAb, anti-HCV Ab, total anti-HDV Ab(for HBsAg positive) and HIV p24 Ag or anti-HIV Ab (confirmed by molecular biology for hepatitis and Western Blot for HIV) will inform respectively on the HBV, HCV, HDV and HIV infection status.

DETAILED DESCRIPTION:
HBV, HCV and HDV are viruses with parenteral, sexual and mother-to-child transmission, associated with high morbidity and mortality. They are responsible for the majority of hepato cellular carcinoma. More than 1.4 million people die each year of complications associated with these infections. Most people do not know their chronic viral hepatitis status which leads to frequent late stage diagnosis of the disease. Treatments allow viral control or suppression of HBV and HCV. The knowledge of the status can reduce transmission,early effective treatment and avoid or delay late complications. In South America, the prevalence of HBV varies widely but is high (> 8%) in the Amazon basin. In some areas a third of HBsAg carriers are also infected with HDV, a major co morbidity factor. French Guiana and Suriname are part of the Amazon biome and are populated by a mosaic of communities. The few available data suggest high variability in hepatitis B and C prevalence in the different communities. The Maroni River is inhabited by Maroon (descendants of slaves of African origin who escaped from Surinamese plantations) and Amerindian communities (indigenous). Reliable data prevalence of HBV, HCV and HIV are lacking in these remote, mobile and vulnerable populations. The infection risk is high, due to low vaccination coverage against HBV, low screening rate and delayed access to care and treatment. There are no data on HDV in this region. In terms of public health, it is of great importance to explore the epidemic of viral hepatitis in the Maroni population pool because the lack of data is an obstacle to the planning of adapted and efficient health interventions.

This multicenter, cross-sectional, population-based study will include 2500 adults in the health care centers / missions located on the 2 sides of the Maroni River. All major inhabitants of the river may participate, after an extensive communication campaign. After signing the informed consent and pre-test counseling, capillary blood will be collected on blotting paper. Participants will be interviewed on infection risk factors. Positivity for HBsAg, total anti-HBcAb, anti-HCV Ab, total anti-HDV Ab(for HBsAg positive) and HIV p24 Ag or anti-HIV Ab (confirmed by molecular biology for hepatitis and Western Blot for HIV) will inform respectively on the HBV, HCV, HDV and HIV infection status. Positive participants will be analyzed in molecular biology (viral load and genotyping). The results will be provided individually and confidentially to participants; positive patients will receive standard care following national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planning to stay on the Maroni river for at least 2 months after inclusion
* Signed informed consent

Exclusion Criteria:

* Consent withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General adult population living along the Maroni River in French Guiana and Suriname, upstream from Apatou. All adults (men and women) 18 years or older of both sexes will be able to participate in the study, in French Guiana and Suriname. Participation will be based on volunteering and signing informed consent. The acceptability and diversity of recruitment will be improved by seeking community support through community leaders and local associations and through appropriate communication (radio spots, posters in health centers and public establishments) before the survey.
Sampling Method: Non-Probability Sample
Enrollment: 2289 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Current active HBV infection | Through study completion, an average of 1 year
  Current active HBV infection determined by HBs Ag positivity
HBV infection carrier status | Through study completion, an average of 1 year
  Acute hepatitis B, chronic active hepatitis B, possible inactive chronic hepatitis B and resolved hepatitis B, determined by HBs Ag and total anti-HBcAb and if HBs Ag is positive by Anti-HBcIgM, HBV DNA and HBe Ag
HCV infection | Through study completion, an average of 1 year
  Anti-HCV Ab positivity confirmed by detection of HCV RNA
HDV infection | Through study completion, an average of 1 year
  Positivity for anti-HDV total Ab (on HBsAg positive samples only) and confirmation by detection of HDV RN
HIV infection | Through study completion, an average of 1 year
  Positive HIV p24 antigen and/or HIV antibodies (fourth-generation combined EIA), confirmed by HIV Ab positivity using Western-blot

SECONDARY OUTCOMES:
Questionnaire | At Enrollment visit
  To describe social and demographic characteristics of infected people and to identify specific risk factors (determinants) associated with HBV, HCV and HIV infection like unsafe sex practices (early sexual initiation, multiple sex partners, not using a condom, traumatic sexual practices, STDs), body modifications (tattoo, piercing, scarifications or bouglous) performed with unsterile equipment, previous blood transfusion or dialysis, sharing personal hygiene equipment like tooth-brush, razor or nail clipper. This will be analyzed using the responses to the questionnaire.
HBV, HCV and HDV genotyping and phylogenetics | Through study completion, an average of 1 year
  Viral sequences will be used for Bayesian analysis of phylogeny and phylogeography. Most recent common ancestor, spreading, risk factors and geographical association will be analyzed for all genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu NACHER, MD, PhD, Study Director — Centre Hospitalier de Cayenne
Locations (2):
- General Hospital of Cayenne, Cayenne, French Guiana
- Foundation for Scientific Research Suriname (SWOS), Paramaribo, Suriname

IPD SHARING:
Plan to Share IPD: No